CLINICAL TRIAL: NCT02701972
Title: Evaluation of Safety and Efficacy of the Basal Annuloplasty of the Cardia Externally (BACE™) [Basal Annuloplasty of the Cardia Externally] Device in the Treatment of Functional Mitral Valve Regurgitation [FMR]
Brief Title: Evaluation of Safety and Efficacy of the BACE™ Device in the Treatment of Functional Mitral Valve Regurgitation [FMR
Acronym: BACE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Phoenix Cardiac Devices, Inc. (Industry)
Collaborators: Toronto General Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BACE CT003
Record Dates: First submitted 2016-02-17; First posted 2016-03-08 (Estimated); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Functional Mitral Regurgitation

STUDY DESIGN:
Intervention Model Description: BACE device implant
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Control and Test (Experimental): Pre-implantation and Post-implantation of BACE device
  Interventions: Device: BACE Device

INTERVENTIONS:
Device: BACE Device — Implanted BACE device

SUMMARY:
The preclinical and clinical evidence of safety and efficacy with the BACE device (concept and feasibility) paved the way for the evaluation of the BACE device in this prospective, multi-center, single-arm, self-controlled study for safety and efficacy in the treatment of functional MR in a maximum of 60 adult subjects.

The primary efficacy endpoint will be reduction of MR grade to 1+ or less from the baseline MR grade through the 6 month study period. Primary safety endpoint will be freedom from major device and surgery-related adverse events for the duration of the 6 month follow up period. Patients will be followed up to two years.

DETAILED DESCRIPTION:
The primary objective of this study is to assess the safety and efficacy of the BACE device for the treatment of FMR.

Secondary objective is to assess the ease of deployment of the BACE device Study Population: Since this study is to assess the safety and efficacy of a new device, with no control arm or comparator, the number of subjects enrolled will be a maximum of 60.

Approximately 8-10 sites are expected to be included in the study. The subject population is adults of 18 to 80 years of age, either gender, with FMR as specified in the inclusion and exclusion criteria.

ELIGIBILITY:
Inclusion Criteria:

* Functional Mitral Valve Regurgitation (FMR) of moderate to severe grade (2 to 4 as per the American College of Cardiology and American Heart Association 2006 Classification of Mitral regurgitation evaluation)
* Symptomatic- NYHA Class II to IV
* Left Ventricular Ejection Fraction (LVEF) 25%-50%
* Normal mitral valve leaflets without any abnormalities and damage
* Subject is willing and available to return for study follow-up
* Surgical approach is the treatment option
* Ability of the subject or legal representative to understand and provide signed consent for participating in the study

Exclusion Criteria:

* Known hypersensitivity or allergy to the device materials
* History or presence of rheumatic heart disease
* Structural abnormality of the mitral valve (e.g. flail leaflets, ruptured or elongated chordae, prolapsed valve, perforated valve leaflets)
* Severe pulmonary hypertension, defined by pulmonary artery systolic (PAS) pressure greater than or equal to 60 mm Hg
* Grade 4 diastolic dysfunction of left ventricle on ECHO, with no change by hemodynamic maneuvers.
* ST segment [of an electrocardiogram] (ST) segment elevation myocardial infarction [MI] within 30 days of enrollment in the study; non ST segment elevation Myocardial Infarction (MI) within 7days of enrollment in the study
* Currently enrolled in another investigational drug or device study
* Subjects with intra-operative [correlate to pre-op measurement end diastolic dimension] heart circumference outside of offered BACE device size ranges [21 to 41 cm]
* Previous mitral valve surgery or other previous cardiac surgery that would preclude proper placement of the BACE
* Abnormal coronary or cardiac anatomy such that the device could not be placed without interfering with those anatomical structures
* Abnormalities in the mitral valve leaflets that would necessitate mitral valve reconstruction or replacement
* Prior Coronary Artery Bypass Graft (CABG) surgery
* Acute active infection
* Active peptic ulcer
* History of IV drug abuse
* Chronic renal failure requiring dialysis
* Creatinine > 2.5 mg/dl
* Open chest surgery contraindication [e.g., acute respiratory distress, endocarditis, myocarditis, pericarditis]
* Immune suppression therapy including corticosteroids
* Subjects with chronic connective tissue disease
* Investigator judgment that body habitus or sternal anatomy precludes pericardial access
* Females who are pregnant or lactating
* Life expectancy of < 12 months due to conditions other than cardiac status

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2016-03; Primary Completion 2021-06-30 (Estimated); Study Completion 2021-09-30 (Estimated)

PRIMARY OUTCOMES:
Reduction in MR grade to MR grade 1+ or less | Two years
  Reduction in Mitral Valve Regurgitation (MR) grade to MR grade 1+ or less after the implantation of the BACE Device as measured by echocardiography.

SECONDARY OUTCOMES:
Durability of or improvement in MR grade over the follow-up period as measured by echocardiography; profiles of the grades in MR based on ECHO at each time point will be plotted for each subject with description of individual percentage change | Two years
  Durability of or improvement in MR grade over the follow-up period as measured by echocardiography
Improvement in cardiac functionality as assessed by the NYHA functional class | Two years
  Improvement in cardiac functionality as assessed by the New York Heart Association (NYHA) functional class
Improvement in cardiac functionality as assessed by the 6-minute walk | Two years
  Improvement in cardiac functionality as assessed by the 6-minute walk
Improvement in cardiac functionality | Two years
  Improvement in cardiac functionality as assessed by the Minnesota Living with Heart Failure questionnaire
All device and surgery-related averse events | Two years
  All device and surgery-related averse events (listed above) and other adverse events over the course of the study will be tabulated

CONTACTS AND LOCATIONS:
Overall Officials: Vivek Rao, MD PhD, Principal Investigator — Toronto General Hospital

IPD SHARING:
Plan to Share IPD: No